CLINICAL TRIAL: NCT06443788
Title: Trans-perineal Ultrasound in Assessment of Preterm Pre-labor Rupture of Membranes Compared to Speculum Examination: Accuracy Study
Brief Title: Trans-perineal Ultrasound in Assessment of PPROMs
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Maya Abdelrazek, Lecturer in Obstetrics and Gynecology, Ain Shams University
Other Study IDs: MS 715/2023
Record Dates: First submitted 2024-05-27; First posted 2024-06-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: PPROM; Preterm Premature Rupture of Membrane
Keywords: transperineal ultrasound; speculum exmaination; PPROM
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women with history suggestive of PPROMs between 24 to 37 weeks' gestation: Evaluation of amniotic fluid pooling via transperineal ultrasonography will be performed. Images will be captured in sagittal and transverse planes. Sagittal plane images will be captured with ultrasound probe placed in between labia major, parallel to their long axis. Transverse plane images will be captured with ultrasound probe placed on posterior fourchette, parallel to the plane of posterior.
  Images will be evaluated for appearance of accumulated hypoechogenic fluid around cervix. Whenever collection is spotted, three largest dimensions of fluid will be measured (length, width, depth).
  Fluid accumulations around the cervix that are clearly demarcated from surrounding tissues were considered positive.
  Cervical length detected . Presenting part and cord prolapse
  Interventions: Diagnostic Test: transperineal ultrasound

INTERVENTIONS:
Diagnostic Test: transperineal ultrasound — The following measurement will be recorded:
  1. Amniotic fluid pooling assessment will be performed in sagittal and transverse planes. ,
     * Images will be evaluated for appearance of accumulated hypoechogenic fluid around cervix. Whenever collection is spotted, three largest dimensions of fluid will be measured (length, width, depth).
     * Fluid accumulations around the cervix that are clearly demarcated from surrounding tissues will be considered positive.
  2. Cervical length: it will be measured between the internal os point to the external os point below. Cervical dilatation will be measured in a transverse plane from inner to inner.
  3. Presence of fetal part prolapse and/or cord prolapse

SUMMARY:
Accurate and timely diagnosis of preterm pre-labor rupture of membranes (PPROM) is important to prevent adverse maternal and fetal outcomes. Following a history of PPROM, physical examination should be performed in a way that minimizes the risk of infection using a speculum. This is important to confirm the diagnosis by visualizing the amniotic fluid passing from the cervical canal or pooling in the vagina. In addition to examining the cervix to assess its dilatation and effacement and look for umbilical cord prolapse or fetal prolapse. However, Pelvic exam is one of the most common anxiety provoking medical procedures that's why this study aims at using the transperineal ultrasound as a non-invasive, accurate, cost effective, applicable and readily available tool in assessment of PPROM with less patient anxiety and fear.

DETAILED DESCRIPTION:
Preterm pre-labor rupture of membranes (PPROM) refers to the disruption of fetal membranes before the beginning of labor, resulting in spontaneous leakage of amniotic fluid. PROM, which occurs prior to 37 weeks of gestation, defined as preterm PROM. The definition is similarly defined by ACOG, NICE, RANZCOG and World Health Organization (WHO).

PROM occurs in approximately 5%-10% of all pregnancies, of which approximately 80% occur at term.

There are numerous risk factors for PPROM, such as intrauterine infection at early gestational age, lower socioeconomic status of pregnant women, inadequate prenatal care and inadequate nutrition during pregnancy, sexually transmitted infections, vaginal bleeding, and smoking during pregnancy.

PPROM is linked to significant maternal and fetal morbidity and mortality. It has been shown to be the cause of 18%-20% and 21.4% of prenatal mortalities and morbidity respectively.

Complications of PPROM for the fetus and newborn consist of prematurity, fetal distress, cord compression, deformation and altered pulmonary development leading to pulmonary hypoplasia and pulmonary hypertension, necrotizing enterocolitis (NEC) and neurologic disorder.

Infectious morbidities in mother, fetus and newborn have been related to both PROM and prolonged rupture of membranes. Maternal complications include intra-amniotic infection, which occurs in 13%-60% of women with PROM, placental abruption, and postpartum endometritis.

Diagnosis of ROM is usually made by observing leakage of the amniotic fluid or by observing the amniotic fluid pooling in the vaginal vault.A golden standard method has not yet been defined in PROM. Diagnostic tests should be used when the diagnosis is not certain following history, examination with sterile speculum and ultrasonography evaluation. Among biochemical tests, PAMG-1 and IGFBP-1 have the features of being easily applicable tests. PAMG-1 comes into prominence with its high sensitivity and specificity. Results of tests used in PROM diagnosis must be supported by clinical findings But in Low resource settings may not have access to some tests due to their cost.

In practice, most complaints of fluid leakage are not due to membrane rupture. However, a complaint of fluid leakage warrants at least a speculum examination to check for amniotic fluid pooling. Speculum examinations are invasive and performing a speculum examination on a patient with the complaint of fluid leakage may be of no consequence when PPROM is ruled out. However, speculum examinations association with the latency periods in PPROM cases is not known and sterile vaginal examinations have been proven to shorten latency periods.

Speculum examination and digital vaginal examination are both similarly invasive in nature, and it may be possible speculum examinations can shorten latency periods as well. Women commonly experience anxiety and fear before and during a pelvic examination. Anxiety or fear has been reported in 21%- 64% of women. Additional studies have reported women experiencing embarrassment of up to 52%, anxiety in 21%-49% and pain in 22%-68%.

The hypothesis of this study is that transperineal ultrasound can be an accurate exam for diagnosis of PPROM and assess of cervical length, effacement and presenting parts in addition to umbilical cord prolapse with less patients anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with history suggestive of preterm prelabor rupture of membranes (PPROM):

  * Sudden gush of fluid per vagina or.
  * Continuous leakage of fluid per vagina or.
  * Feeling wet or.
  * Feeling inability to stop urinating.
* 24 to 37 weeks' gestation.

Exclusion Criteria:

* • Women in active labor (uterine contraction with cervical dilatation more than or equal to 5 cm).

  * Women with vaginal bleeding.
  * Vulvovaginitis (vaginal discharge).
  * Cervical cerclage in place.
  * Intrauterine fetal demise (IUFD).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with a history suggestive of preterm prelabor rupture of membranes (PPROM) presenting to the emergency ward or the outpatient clinic at Ain Shams University Maternity Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Accuracy in diagnosis of PPROM by trans-perineal ultrasound | at time of diagnosis (24 to 37 weeks' gestation)
  Images by ultrasound will be evaluated for appearance of accumulated hypoechogenic fluid around cervix. Whenever collection is spotted, three largest dimensions of fluid will be measured (length, width, depth) comparing it to speculum examination by observing amniotic fluid leaking through the cervix or pooling of amniotic fluid in posterior vaginal vault

SECONDARY OUTCOMES:
assessment of cervical length and dilatation by ultrasound (objective) in mm. | at time of diagnosis (24 to 37 weeks' gestation)
  comapred to speculum examination (subjective)
assessment of fetal parts or cord prolapse by ultrasound | at time of diagnosis (24 to 37 weeks' gestation)
  compared to visualization by speculum (visualizing any fetal part or cord prolapsiing from the cervix)
assessment of patients' anxiety (Tolerability to the examination) | at time of diagnosis (24 to 37 weeks' gestation)
  using State-Trait Anxiety Inventory (STAI). 1 = not at all / almost never, 2 = somewhat/sometimes, 3 = moderately so / often, and 4 = very much so / almost always

CONTACTS AND LOCATIONS:
Overall Officials: Maya M. Abdelrazek, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No